CLINICAL TRIAL: NCT01351467
Title: Ongoing, Web-Based Genome-Wide Association Studies for Targeted Disease Initiatives
Brief Title: Web-based Genetic Research on Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: 23andMe, Inc. (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); The Parkinson's Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 23andMe_PD001
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's; genetic; online; GWAS; genome wide association
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples are collected for DNA analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinson's disease patients: People diagnosed with Parkinson's disease by a physician

SUMMARY:
The purpose of this study is to examine how genes and environment affect risk for Parkinson's disease.

DETAILED DESCRIPTION:
23andMe has created a web-based Parkinson's research initiative to understand the genetic associations found between Parkinson's patients' DNA and their disease. To learn more, visit: https://www.23andme.com/pd/. You can participate in this research initiative without leaving home. If you are eligible to participate, we will send you an in-home 23andMe DNA kit at no cost. We will ask you short online surveys (15-20) about your Parkinson's journey, symptoms, and response to treatment. Enrollment is on-going and open to individuals who have been diagnosed with Parkinson's disease and are residents of the U.S. Participants receive access to ancestry information and uninterpreted genetic data. Participants will also receive regular updates on our research efforts and findings.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease by a physician

Exclusion Criteria:

* diagnoses other than Parkinson's, including:
* progressive supranuclear palsy (PSP)
* multiple system atrophy (MSA)
* Shy-Drager syndrome
* spinal cerebella ataxia (SCA)
* atypical parkinsonism
* parkinsonism due to medications, drug-induced parkinsonism
* vascular parkinsonism
* frontotemporal dementia with parkinsonism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 13576 (Actual)
Dates: Start 2009-04; Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Saliva DNA test and online surveys with questions about Parkinson's disease experience, symptoms and response to treatment | Intermittent surveys every 6 months for up to 24 months
  We want to learn how genes and environment could play role in Parkinson's disease risk and progression

CONTACTS AND LOCATIONS:
Locations (1):
- Www.23Andme.Com/Pd, Mountain View, California, United States

REFERENCES:
- [Result] Do CB, Tung JY, Dorfman E, Kiefer AK, Drabant EM, Francke U, Mountain JL, Goldman SM, Tanner CM, Langston JW, Wojcicki A, Eriksson N. Web-based genome-wide association study identifies two novel loci and a substantial genetic component for Parkinson's disease. PLoS Genet. 2011 Jun;7(6):e1002141. doi: 10.1371/journal.pgen.1002141. Epub 2011 Jun 23. PMID 21738487
- [Result] Lill CM, Roehr JT, McQueen MB, Kavvoura FK, Bagade S, Schjeide BM, Schjeide LM, Meissner E, Zauft U, Allen NC, Liu T, Schilling M, Anderson KJ, Beecham G, Berg D, Biernacka JM, Brice A, DeStefano AL, Do CB, Eriksson N, Factor SA, Farrer MJ, Foroud T, Gasser T, Hamza T, Hardy JA, Heutink P, Hill-Burns EM, Klein C, Latourelle JC, Maraganore DM, Martin ER, Martinez M, Myers RH, Nalls MA, Pankratz N, Payami H, Satake W, Scott WK, Sharma M, Singleton AB, Stefansson K, Toda T, Tung JY, Vance J, Wood NW, Zabetian CP; 23andMe Genetic Epidemiology of Parkinson's Disease Consortium; International Parkinson's Disease Genomics Consortium; Parkinson's Disease GWAS Consortium; Wellcome Trust Case Control Consortium 2); Young P, Tanzi RE, Khoury MJ, Zipp F, Lehrach H, Ioannidis JP, Bertram L. Comprehensive research synopsis and systematic meta-analyses in Parkinson's disease genetics: The PDGene database. PLoS Genet. 2012;8(3):e1002548. doi: 10.1371/journal.pgen.1002548. Epub 2012 Mar 15. PMID 22438815
- [Result] Pichler I, Del Greco M F, Gogele M, Lill CM, Bertram L, Do CB, Eriksson N, Foroud T, Myers RH; PD GWAS Consortium; Nalls M, Keller MF; International Parkinson's Disease Genomics Consortium; Wellcome Trust Case Control Consortium 2; Benyamin B, Whitfield JB; Genetics of Iron Status Consortium; Pramstaller PP, Hicks AA, Thompson JR, Minelli C. Serum iron levels and the risk of Parkinson disease: a Mendelian randomization study. PLoS Med. 2013;10(6):e1001462. doi: 10.1371/journal.pmed.1001462. Epub 2013 Jun 4. PMID 23750121
- [Result] Nalls MA, Pankratz N, Lill CM, Do CB, Hernandez DG, Saad M, DeStefano AL, Kara E, Bras J, Sharma M, Schulte C, Keller MF, Arepalli S, Letson C, Edsall C, Stefansson H, Liu X, Pliner H, Lee JH, Cheng R; International Parkinson's Disease Genomics Consortium (IPDGC); Parkinson's Study Group (PSG) Parkinson's Research: The Organized GENetics Initiative (PROGENI); 23andMe; GenePD; NeuroGenetics Research Consortium (NGRC); Hussman Institute of Human Genomics (HIHG); Ashkenazi Jewish Dataset Investigator; Cohorts for Health and Aging Research in Genetic Epidemiology (CHARGE); North American Brain Expression Consortium (NABEC); United Kingdom Brain Expression Consortium (UKBEC); Greek Parkinson's Disease Consortium; Alzheimer Genetic Analysis Group; Ikram MA, Ioannidis JP, Hadjigeorgiou GM, Bis JC, Martinez M, Perlmutter JS, Goate A, Marder K, Fiske B, Sutherland M, Xiromerisiou G, Myers RH, Clark LN, Stefansson K, Hardy JA, Heutink P, Chen H, Wood NW, Houlden H, Payami H, Brice A, Scott WK, Gasser T, Bertram L, Eriksson N, Foroud T, Singleton AB. Large-scale meta-analysis of genome-wide association data identifies six new risk loci for Parkinson's disease. Nat Genet. 2014 Sep;46(9):989-93. doi: 10.1038/ng.3043. Epub 2014 Jul 27. PMID 25064009
- See also: Click here for more information about this study: Web-based Genetic Research on Parkinson's Disease — https://www.23andme.com/pd